CLINICAL TRIAL: NCT03161132
Title: Multicentric Single Arm Phase II Clinical Trial, to Evaluate Safety and Efficacy of the Combination of Olaparib and PLD for Platinum Resistant Ovarian Primary Peritoneal Carcinoma, and Fallopian Tube Cancer Patients.
Brief Title: Resistant Ovarian Cancer, Olaparib and Liposomal Doxorubicin
Acronym: ROLANDO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICO-1601; 2016-004850-14 (EudraCT Number)
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Advanced Ovarian Cancer
MeSH Terms: interventions — olaparib; liposomal doxorubicin; 1-dodecylpyridoxal

STUDY DESIGN:
Intervention Model Description: Multicentric
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olaparib 300mg (Experimental): Olaparib bid orally at 300 mg (tablet formulation) continuously, combined with chemotherapy with Pegylated Liposomal Doxorubicin (up to 6 cycles), then, as monotherapy at the same dose and frequency (300mg bid orally) until progression of disease or unaccepted toxicity.
  Interventions: Drug: Olaparib
- Pegylated Liposomal Doxorubicin (PLD) (Other): PLD 40mg/m2 every 28 days intravenous for up to 6 cycles. This treatment will be combined with Olaparib (as described earlier).
  Interventions: Drug: Pegylated Liposomal Doxorubicin

INTERVENTIONS:
Drug: Olaparib — Combination of continous olaparib 300mg for oral administration plus Pegylated Liposomal Doxorubicin (PLD), followed by maintenance treatment further described.
  Other Names: Lynparza
  Arms: Olaparib 300mg
Drug: Pegylated Liposomal Doxorubicin — PLD 40mg/m2 every 28 days intravenous
  Other Names: PLD
  Arms: Pegylated Liposomal Doxorubicin (PLD)

SUMMARY:
Impact of the combination of Olaparib and Pegylated Liposomal Doxorubicin on improvement of progression-free survival at 6 months in patients with platinum resistant advanced ovarian cancer.

DETAILED DESCRIPTION:
The combination of Poly (ADP-ribose) polymerase (PARP) inhibitors with PLD may provide a synergistic effect in patients with advanced ovarian cancer, especially those with Homologous recombination deficiency (HRD), because of the decreased ability to repair chemotherapy-induced DNA damage. Preclinical studies with PARP inhibitors have shown potentiation of the cytotoxic effects of chemotherapeutic agents and a recent phase I study has shown the tolerability of the combination and efficacy in recurrent ovarian cancer. In this study, encouraging efficacy results were seen in ovarian cancer patients and were not limited by Germline BRCA1/2 (gBRCA) Mutations status or sensitivity to platinum therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures. Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and those obtained prior to signing of informed consent may be utilized for screening or for baseline purposes provided these procedures are conducted as specified in the protocol.
* Patients with histological or cytological confirmed high grade serous or endometrioid epithelial ovarian cancer, primary peritoneal carcinoma, fallopian tube cancer and resistant platinum relapse with no prior treatment with PLD for their resistant relapse. Previous treatment with PLD is allowed as long as it was part of one platinum based regimen and the treatment was finalized at least six months previously to inclusion in this trial.
* Patients must have platinum-resistant disease, defined as progression within <6 months from completion of at least 4 cycles of platinum and up to 3 prior chemotherapy regimens. Patients should have documented treatment-free interval of ≥6 months following 1st chemotherapy regimen received. Patients with a deleterious mutation in BRCA are eligible in any case with a resistant relapse including primary resistant relapse.
* Have measurable disease as defined by RECIST v1.1 Criteria. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Female patients with > 18 years of age.
* Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below: Haemoglobin ≥ 10.0 g/dL; Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; No features suggestive of Myelodysplastic Syndrome/Acute Myeloid Leukemia on peripheral blood smear; White blood cells (WBC) > 3x109/L; Platelet count ≥ 100 x 109/L; Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN); aspartate aminotransferase (AST/SGOT)/Alaninotransferase (ALT/SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN.
* Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min. PLD is metabolised by the liver and excreted in the bile. Population pharmacokinetic data (in the range of creatinine clearance tested of 30-156 ml/min) demonstrate that PLD clearance is not influenced by renal function. No pharmacokinetic data are available in patients with creatinine clearance of less than 30 ml/min.
* Patients must have a life expectancy ≥ 16 weeks.
* Evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1 Postmenopausal is defined as: Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments; luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the postmenopausal range for women under 50; Radiation-induced oophorectomy with last menses >1 year ago; Chemotherapy-induced menopause with >1 year interval since last menses; or surgical sterilisation (bilateral oophorectomy or hysterectomy).
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
* Left Ventricular Ejection Fraction (LVEF) ≥ 50%.

Exclusion Criteria:

* Platinum-refractory disease (progression during previous platinum therapy).
* Involvement in the planning and/or conduct of the study (applies to both Sponsor staff and/or staff at the study site).
* Previous enrolment in the present study.
* Participation in another clinical study with an investigational product during the last 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study treatment.
* Any previous treatment with a PARP inhibitor, including olaparib.
* Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥5 years.
* Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment with study drug.
* Concomitant use of known CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir.
* Persistent toxicities (>=CTCAE grade 2) with the exception of alopecia, caused by previous cancer therapy.
* Resting ECG with corrected QT interval (QTc) >470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
* Blood transfusions within 28 days prior to study entry.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia.
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 28 days prior to treatment.
* Major surgery within 14 days of starting study treatment and patients must have recovered from any effects of any major surgery.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, unstable spinal cord compression (untreated and unstable for at least 28 days prior to study entry), superior vena cava syndrome, extensive bilateral lung disease on high-resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Breast feeding women.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving antiviral therapy.
* Patients with known active hepatic disease (i.e., Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Patients with a known hypersensitivity to the combination/comparator agent
* Patients with uncontrolled seizures.
* Previous allogeneic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival | 6 months
  Proportion of pacients with no progression of disease at 6 months after start of treatment with Olaparib plus PLD

SECONDARY OUTCOMES:
Objective Response Rate | 20 months
  Proportion of patients with tumor size reduction. Response duration is measured from the time of initial response until documented tumor progression. The Objective Response Rate (ORR) is defined as the sum of partial responses plus complete responses according to RECIST 1.1.
Disease Control Rate | 20 months
  Proportion of patients who have achieved complete response, partial response and stable disease of 8 or more months according to RECIST 1.1
Response to treatment Rate according CA-125 levels | 20 months
  Proportion of patients who have achieved a response according to CA-125: and it has occurred if there is at least a 50% reduction in CA-125 levels from a pretreatment sample.
Progression-free survival | 20 months
  Time from the date of the first dose of study treatment to the date of objective disease progression or death (in the absence of progression) regardless of whether the subject withdraws from study treatment or receives another anti-cancer therapy prior to progression.
Overall survival | 20 months
  Time from inclusion until death of any cause.
Health related quality of life | 20 months
  Change in patient's quality of life during the study, using the self-reported European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) (EORTC QLQ-C30) and the EORTC ovarian cancer module (EORTC-OV-28). Both scores will be combined to report a final outcome.
Activity of tumor based on the growth modulation index (GMI) | 20 months
  The GMI is the ratio of time to progression with the nth line (TTP(n)) of therapy to the TTP(n)(-1) with the n-1th line. GMI >1.33 is considered as a sign of activity in phase II trials.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 20 months
  Frequency, nature and number of patients developing adverse events throughout follow up
DNA damage | 20 months
  BRCA pathway and defects in homologous recombination repair (HRR) Phosphorylation of γH2AX as a marker of DNA damage.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Pérez-Fidalgo, M.D., Ph.D., Principal Investigator — University of Valencia, Hospital Clinico Universitario de Valencia
Locations (8):
- Spain (8):
  - Corporación Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Son Llatzer, Palma de Mallorca, Mallorca
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez-Fidalgo JA, Iglesias M, Bohn U, Calvo E, Garcia Y, Guerra E, Manso L, Santaballa A, Gonzalez-Martin A. GEICO1601-ROLANDO: a multicentric single arm Phase II clinical trial to evaluate the combination of olaparib and pegylated liposomal doxorubicin for platinum-resistant ovarian cancer. Future Sci OA. 2019 Jan 10;5(2):FSO370. doi: 10.4155/fsoa-2018-0107. eCollection 2019 Feb. PMID 30820349
- [Result] Perez-Fidalgo JA, Cortes A, Guerra E, Garcia Y, Iglesias M, Bohn Sarmiento U, Calvo Garcia E, Manso Sanchez L, Santaballa A, Oaknin A, Redondo A, Rubio MJ, Gonzalez-Martin A. Olaparib in combination with pegylated liposomal doxorubicin for platinum-resistant ovarian cancer regardless of BRCA status: a GEICO phase II trial (ROLANDO study). ESMO Open. 2021 Aug;6(4):100212. doi: 10.1016/j.esmoop.2021.100212. Epub 2021 Jul 27. PMID 34329939